CLINICAL TRIAL: NCT01318252
Title: AL-54478 Proof of Concept Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-10-080
Record Dates: First submitted 2011-03-16; First posted 2011-03-18 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Open-angle Glaucoma (OAG); Ocular Hypertension (OHT)
Keywords: Elevated IOP
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AL-54478 (Experimental): AL-54478 0.005%, single dose, followed 7 days later with 14 days of once daily dosing
  Interventions: Drug: AL-54478 0.005%
- Latanoprost (Active Comparator): Latanoprost 0.005%, single dose, followed 7 days later with 14 days of once daily dosing
  Interventions: Drug: Latanoprost 0.005%
- Vehicle (Placebo Comparator): AL-54478 Vehicle, single dose, followed 7 days later with 14 days of once daily dosing
  Interventions: Drug: AL-54478 Vehicle

INTERVENTIONS:
Drug: AL-54478 0.005%
  Arms: AL-54478
Drug: Latanoprost 0.005%
  Arms: Latanoprost
Drug: AL-54478 Vehicle — Inactive ingredients used as a placebo comparator
  Arms: Vehicle

SUMMARY:
The purpose of this study is to assess the safety and efficacy of AL-54478 0.005% compared with Latanoprost 0.005% and AL-54478 Vehicle in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with either OAG or OHT.
* Patients who are able to comply with the scheduled visits.
* Patients who have had a physical exam within 6 months of the Screening Visit.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Females of childbearing potential who meet any 1 of the following conditions: a) Currently pregnant; b) Positive urine pregnancy test; c)Intend to become pregnant; d) Breast feeding; e) Not using highly effective birth control measures.
* Patients with extreme narrow angle with complete or partial closure.
* Patients with a cup to disc ratio more than 0.8.
* Patients with a severe central visual field loss in either eye.
* Patients with chronic or recurrent inflammatory eye disease or acute ocular infection or inflammation.
* Patients who have had ocular trauma within the past 6 months or have had intraocular surgery within the past 6 months or have had ocular laser surgery within the past 3 months.
* Patients with best-correct visual acuity less than 20/80.
* Patients who have had ocular infection or inflammation within the past 3 months.
* Patients who have clinically relevant progressive retinal disease.
* Patients who have severe illness or conditions.
* Patients who have hypersensitivity to a prostaglandin analogu.e
* Patients who are unable to safely discontinue all IOP-lowering medications during washout.
* Patients who are currently on therapy with another investigational agent within 30 days prior to the Screening Visit.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
24-hour Area Under the Curve (AUC) for IOP Change from Baseline after 14 Days of Once Daily Dosing | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Ravaughn Williams, Study Director — Alcon Research